CLINICAL TRIAL: NCT05330728
Title: Comparison of the Effects of Abdominal Massage and Kinesio Taping in Women With Chronic Constipation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, seyda toprak celenay, associate professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/04/10
Record Dates: First submitted 2022-04-09; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Suggestion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Massage group (Experimental): Suggestions for lifestyle changes + abdominal massage will be performed.
  Interventions: Other: Suggestions for lifestyle changes+ Abdominal massage
- Taping group (Active Comparator): Suggestions for Lifestyle Changes + Kinesio taping will be performed.
  Interventions: Other: Suggestions for lifestyle changes+ Kinesio taping
- Control group (Other): Suggestions for lifestyle changes will be performed.
  Interventions: Other: Suggestions for lifestyle changes

INTERVENTIONS:
Other: Suggestions for lifestyle changes+ Abdominal massage — Suggestions for lifestyle changes+ abdominal massage will be applied. Suggestions including regular and balanced diet, fluid consumption, regular walking and abdominal exercises and correct toilet habits will be given once. Abdominal massage will be applied 3 times a week for 4 weeks.
  Arms: Massage group
Other: Suggestions for lifestyle changes+ Kinesio taping — Suggestions including regular and balanced diet, fluid consumption, regular walking and abdominal exercises and correct toilet habits will be given once. Kinesio taping will be applied 3 times a week for 4 weeks.
  Arms: Taping group
Other: Suggestions for lifestyle changes — Suggestions including regular and balanced diet, fluid consumption, regular walking and abdominal exercises and correct toilet habits will be given once.
  Arms: Control group

SUMMARY:
The aim of this study is to compare the effects of abdominal massage and kinesio taping on constipation severity, quality of life, bowel habits and perception of recovery in women with chronic constipation.

DETAILED DESCRIPTION:
Constipation is not a disease but a subjective symptom characterized by inadequate defecation, the definition of which varies from person to person. It is known that abdominal massage, which is one of the physiotherapy approaches, reduces the severity of gastrointestinal symptoms and increases bowel movements. Kinesio taping applied for constipation can also increase bowel movement, increase the frequency of defecation and decrease the duration of defecation. However, there is a need for studies comparing the effects of these two different applications.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age
* Having been diagnosed with chronic constipation according to the Rome 4 diagnostic criteria by a gastroenterologist
* Being volunteer

Exclusion Criteria:

* Concomitant colon or gastrointestinal problems
* Body mass index >35 kg/m2
* Those who have difficulty defecating, those with anorectal dyssynergia
* Being pregnant
* Having neurological, metabolic and/or malignant disease
* Having an open wound, mass, infection and/or hernia in the area to be massaged
* Having abdominal surgery or abdominal radiotherapy in the last 1 year
* Having a mental problem that prevents cooperation
* Taking laxative therapy at least 4 weeks before participating in the study
* To have received physiotherapy and rehabilitation applications related to constipation in the last 1 year

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2022-08-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Constipation severity | change from baseline at 4 weeks
  Constipation severity will be evaluated with Constipation Severity Scale. According to constipation severity scale, women's defecation frequency, intensity and difficulty/difficulty during defecation will be determined. The scale, which includes sixteen questions, consists of 3 sub-groups: obstructive defecation, colonic inertia and pain. The score that can be obtained from the obstructive defecation subgroup is 0-28, the score that can be obtained from the colonic inertia subgroup is 0-29, and the score that can be obtained from the pain subgroup is between 0-16. The lowest total score that can be obtained from the constipation severity scale is 0, and the highest is 73. As the score obtained from the scale increases, the severity of the symptoms increases.

SECONDARY OUTCOMES:
Life quality | change from baseline at 4 weeks
  Life quality will be evaluated with Constipation Quality of Life Scale. It includes a total of 28 items in 4 subscales: worries and concerns (11 items), physical discomfort (4 items), psychosocial discomfort (8 items), and satisfaction (5 items). Item scores of the five-point Likert-type scale range from 1 to 5. The highest score that can be obtained from the scale is 140, and the lowest score is 28. It is stated that as the scores obtained from the scale increase, the quality of life may also be negatively affected.
Bowel habits | change from baseline at 4 weeks
  Bowel habits will be evaluated with 7-day bowel diary. This diary included items related to frequency of bowel movement, defecation time, feeling of incomplete evacuation, medication use, and changes in food and liquid consumption.
Stool consistency | change from baseline at 4 weeks
  Stool consistency will be assessed using Bristol Stool Scale on a 7-point scale (from 1 to 7) which is a quick and useful indicator of colonic transit time: type 1 = separate hard lumps, like nuts; 2 = sausage shaped but lumpy; 3 = like a sausage or snake, but with cracks on its surface; 4 = like a sausage or snake, smooth and soft; 5 = soft blobs with clear-cut edges; 6 = fluffy pieces with ragged edges, a mushy stool; and 7 = water, no solid pieces.
Perception of recovery | change from baseline at 4 weeks
  Perception of recovery will be evaluated using a 4-point Likert-type scale. Accordingly, women will be asked to choose one of the statements as "worse, same, better or better" regarding the decrease in the severity of constipation when compared before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Principal Investigator — Ankara Yildirim Beyazıt University